CLINICAL TRIAL: NCT05392660
Title: Effect of Upright Position During First Stage of Labour On Labour Outcome: An Evidence Based Approach
Brief Title: Upright Position During First Stage of Labour
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rabab sabry hassen mohamed, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2014
Record Dates: First submitted 2022-05-19; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Effects of Movement
Keywords: First stage of labor; Upright position; Labor outcomes

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Allocation of the women to study or control group was carried out through a person not involved in the study nurses in charge during the shift. This allocation was concealed from person allocating a woman into the trial (nurses)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study arm (Experimental): assumed upright position during first stage of labor
  Interventions: Other: assumed upright position during first stage of labor
- control arm (No Intervention): hospital routine care

INTERVENTIONS:
Other: assumed upright position during first stage of labor — The study group assumed one of upright positions during first stage of labor, defined as walking , sitting, standing, kneeling & squatting positions )
  Arms: study arm

SUMMARY:
There are several physiological advantages for being upright during labour. These include the effect of gravity on the fetus within the uterus; reduced risk of aorto-caval compression this maximizes uterine blood ﬂow to the placenta and fetus during labour and more efficient contractions which lead to shorter first and second stage of labor. In addition, being upright during labour provide better alignment of the fetus; and increased pelvic outlet when the woman is in squatting and kneeling positions

ELIGIBILITY:
Inclusion Criteria:

* Primipara parturient women who admitted to delivery unit;
* in early active phase of 1st stage of labor (not more than 4cm),
* age between 20-35 years,
* had a single, viable, and full term (≥ 37 weeks),
* with normal fetal heart rate pattern (120-160 b/min),
* fetus in occipto anterior position
* free from medical or obstetrical disorders that may interrupt labor progress

Exclusion Criteria:

* Any women out of inclusion criteria

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2020-03-27 (Actual); Study Completion 2020-03-27 (Actual)

PRIMARY OUTCOMES:
Intensity of labor pain assessed by Visual analogue pain intensity scale | during the procedure
  Assessment of labor pain assessed by VAS (Visual analogue pain intensity scale ).It is a self-reported 10 cm horizontal line which represented the subjective estimation of pain intensity. It comprised 0-10-point numerical scale, No pain (0), Mild pain (< 4), Moderate pain (4-6), Sever pain (7-10).
duration of first stage of labor | during the procedure
  upright position may decrease the duration of first stage of labor

SECONDARY OUTCOMES:
duration of second stage of labor | immediately after intervention
  upright position may decrease the duration of second stage of labor
fetal outcome | during the procedure
  fetal well being through fetal heart rate assessment assessed by CTG (cardio toco graph ) machine
Neonatal outcome | immediately after intervention
  neonatal condition after delivery assessed by a standardized APGAR score tool by allocating scores to five simple criteria Activity (Muscle tone), Pulse (Heart rate), Grimace (reflex irritability) Appearance (Skin color) & Respiratory effort (breathing). A total score (0-3) revealed sever neonatal distress, (4-7) indicated moderate distress & (8-10) indicated absence of difficulty in adjusting to extra uterine live.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of nursing Cairo university, Cairo, Egypt